CLINICAL TRIAL: NCT06339671
Title: Complicanze Post-operatorie e Abitudine Tabagica in Chirurgia Colorettale (Studio PASSAGE). Uno Studio Multicentrico Osservazionale Prospettico e Retrospettivo in Italia
Brief Title: Post-operative Complications and Smoking Habits in Colorectal Surgery
Acronym: PASSAGE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Collaborators: Ospedale San Paolo (Other); Ospedali Riuniti Marche Nord pesaro (Unknown)
Responsible Party: Principal Investigator, Pierpaolo Sileri, Professor, IRCCS Ospedale San Raffaele
Other Study IDs: PASSAGE
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NF (Non fumatori): Non-smoker
- FT (Fumatori di tobacco): Tobacco smokers
- NRT (Nicotine replacement therapy): Nicotine replacement therapy

SUMMARY:
PASSAGE is a national multicenter retrospective and prospective observational cohort study in which patients who will undergo colorectal surgery will be enrolled.

DETAILED DESCRIPTION:
The first part of the study is retrospective and data collection will be done the first 6 months. The enrolled patients will be divided into three groups (FT: tobacco smokers; NRT: nicotine replacement therapy; NF: non-smokers) and the data will be compared between groups to evaluate whether there are statistically significant differences regarding postoperative complications. The NF group will also be divided into patients who have never smoked and patients who have stopped smoking. A further analysis of ex-smoking patients will be performed to evaluate whether the incidence of complications differs from that observed in patients who have never smoked. The second part of the study will be prospective and will last one year. Also in this study the enrolled patients will be divided into three groups (NF group, FT group, and NRT group) and data obtained from all recorded variables will be compared between the groups. The data obtained retrospectively and prospectively will be analyzed together for each group.

The hypothesis of the study is that tobacco smoking plays a significant role in the appearance of postoperative complications. In particular, it is hypothesized that the group of patients taking NRT (defined as the group of NRT patients) has a higher incidence of postoperative complications after colorectal surgery than that observed in the control group of non-smoking (NF) or ex-smoking patients and lower to the group of tobacco smoking patients (FT).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* Patients who have read, understood, accepted and signed the informed consent to the study.
* Patients with benign or malignant colorectal disease.
* Patients undergoing colorectal surgery with any type of approach (open or minimally invasive) in Italy.
* Patients undergoing elective and emergency colorectal surgery.
* Patients NF (non smoker), FT (tobacco smokers), NRT (nicotine replacement therapy). Are considered smokers that patients who have smoked for at least 30 days at the time of surgery

Exclusion Criteria:

* Patients < 18 years old.
* Patients who have not accepted informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone colorectal surgery. Patients who need to undergo colorectal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1527 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of postoperative complications surgery in three groups | 30 days
  Incidence of postoperative complications (new onset) within 30 days from the date of surgery in the three groups of patients (NF, FT, NRT).

SECONDARY OUTCOMES:
Incidence and severity of postoperative complications surgery in NF (non-smokers) group | 30 days
  Incidence of postoperative complications (new onset) within 30 days from the date of surgery in the two groups of NF patients (patients who have never smoked and patients who have stopped smoking).

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Sileri, Prof., Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- Prof. Pierpaolo Sileri, Milan, Italy

REFERENCES:
- [Background] Gaskill CE, Kling CE, Varghese TK Jr, Veenstra DL, Thirlby RC, Flum DR, Alfonso-Cristancho R. Financial benefit of a smoking cessation program prior to elective colorectal surgery. J Surg Res. 2017 Jul;215:183-189. doi: 10.1016/j.jss.2017.03.067. Epub 2017 Apr 7. PMID 28688645
- [Background] Gronkjaer M, Eliasen M, Skov-Ettrup LS, Tolstrup JS, Christiansen AH, Mikkelsen SS, Becker U, Flensborg-Madsen T. Preoperative smoking status and postoperative complications: a systematic review and meta-analysis. Ann Surg. 2014 Jan;259(1):52-71. doi: 10.1097/SLA.0b013e3182911913. PMID 23799418
- [Background] Balla A, Saraceno F, Rullo M, Morales-Conde S, Targarona Soler EM, Di Saverio S, Guerrieri M, Lepiane P, Di Lorenzo N, Adamina M, Alarcon I, Arezzo A, Bollo Rodriguez J, Boni L, Biondo S, Carrano FM, Chand M, Jenkins JT, Davies J, Delgado Rivilla S, Delrio P, Elmore U, Espin-Basany E, Fichera A, Flor Lorente B, Francis N, Gomez Ruiz M, Hahnloser D, Licardie E, Martinez C, Ortenzi M, Panis Y, Pastor Idoate C, Paganini AM, Pera M, Perinotti R, Popowich DA, Rockall T, Rosati R, Sartori A, Scoglio D, Shalaby M, Simo Fernandez V, Smart NJ, Spinelli A, Sylla P, Tanis PJ, Valdes-Hernandez J, Wexner SD, Sileri P. Protective ileostomy creation after anterior resection of the rectum: Shared decision-making or still subjective? Colorectal Dis. 2023 Apr;25(4):647-659. doi: 10.1111/codi.16454. Epub 2022 Dec 28. PMID 36527323
- [Background] Tsai KY, Huang SH, You JF, Tang R, Chiang JM, Yeh CY, Hsieh PS, Tsai WS, Chiang SF, Lai CC. Smoking cessation for less than 10 years remains a risk factor of anastomotic leakage in mid-to-low rectal cancer patients undergoing sphincter-preserving surgery. Langenbecks Arch Surg. 2022 May;407(3):1131-1138. doi: 10.1007/s00423-021-02381-9. Epub 2022 Jan 26. PMID 35079889
- [Background] Silverstein P. Smoking and wound healing. Am J Med. 1992 Jul 15;93(1A):22S-24S. doi: 10.1016/0002-9343(92)90623-j. PMID 1323208
- [Background] Guerif V, Atlan M, Cristofari S. Pathophysiology of nicotine, place of nicotine substitutes and electronic cigarettes in plastic surgery: A review of the literature. Ann Chir Plast Esthet. 2022 Jun;67(3):119-124. doi: 10.1016/j.anplas.2022.05.001. Epub 2022 Jun 4. PMID 35672174
- [Background] Turan A, Mascha EJ, Roberman D, Turner PL, You J, Kurz A, Sessler DI, Saager L. Smoking and perioperative outcomes. Anesthesiology. 2011 Apr;114(4):837-46. doi: 10.1097/ALN.0b013e318210f560. PMID 21372682
- [Background] Shi Y, Warner DO. Surgery as a teachable moment for smoking cessation. Anesthesiology. 2010 Jan;112(1):102-7. doi: 10.1097/ALN.0b013e3181c61cf9. PMID 19996946
- [Background] Parthasarathy M, Greensmith M, Bowers D, Groot-Wassink T. Risk factors for anastomotic leakage after colorectal resection: a retrospective analysis of 17 518 patients. Colorectal Dis. 2017 Mar;19(3):288-298. doi: 10.1111/codi.13476. PMID 27474844
- [Background] Zhang W, Lou Z, Liu Q, Meng R, Gong H, Hao L, Liu P, Sun G, Ma J, Zhang W. Multicenter analysis of risk factors for anastomotic leakage after middle and low rectal cancer resection without diverting stoma: a retrospective study of 319 consecutive patients. Int J Colorectal Dis. 2017 Oct;32(10):1431-1437. doi: 10.1007/s00384-017-2875-8. Epub 2017 Aug 2. PMID 28766076
- [Background] Shahab L, Goniewicz ML, Blount BC, Brown J, McNeill A, Alwis KU, Feng J, Wang L, West R. Nicotine, Carcinogen, and Toxin Exposure in Long-Term E-Cigarette and Nicotine Replacement Therapy Users: A Cross-sectional Study. Ann Intern Med. 2017 Mar 21;166(6):390-400. doi: 10.7326/M16-1107. Epub 2017 Feb 7. PMID 28166548
- [Background] Sun R, Mendez D, Warner KE. Trends in Nicotine Product Use Among US Adolescents, 1999-2020. JAMA Netw Open. 2021 Aug 2;4(8):e2118788. doi: 10.1001/jamanetworkopen.2021.18788. PMID 34432013
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Background] Choe SI, Finley C. Confronting the Negative Impact of Cigarette Smoking on Cancer Surgery. Curr Oncol. 2022 Aug 18;29(8):5869-5874. doi: 10.3390/curroncol29080463. PMID 36005201
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450
- See also: National Academies of Sciences, Engineering, and Medicine. 2018. Public health consequences of e-cigarettes. Accessed March 8, 2023 — https://nap.nationalacademies.org/catalog/24952/public-health-consequences-of-e-cigarettes